CLINICAL TRIAL: NCT05602662
Title: Music as a Complement to Pharmacological Sedation in Ventilator Treated ICU Patients - Prospective Randomized Cross-over Study.
Brief Title: Music as a Complement to Pharmacological Sedation in Ventilator Treated ICU Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad Central Hospital (Other)
Collaborators: University Hospital of Uppsala Sweden (Unknown); University Hospital of Gothenburg Sweden (Unknown); Central Hospital of Gävle, Sweden (Unknown); Central Hospital of Falun Sweden (Unknown); University Hospital of Örebro Sweden (Unknown)
Responsible Party: Principal Investigator, Ragnar Henningsson, Associate Professor, Karlstad Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KarlstadCH2
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Music Therapy
Keywords: Music therapy, Ventilator treated patients, Need of sedation.
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy during mechanical ventilation in the iCU. (Experimental): Headphones with music.
  Interventions: Behavioral: Music
- Comparator (Sham Comparator): Headphones only.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Music therapy during mechanical ventilation

SUMMARY:
Can music theraphy during mechanical ventilation in the ICU, decrease the need of pharmacological sedation? Included patients will listen to music selected by a music therapist via headphones two times one hour during two days. Effects on heart rate, blood pressure, respiratory rate and dosing of pharmacological sedation will be observed. 100 patients will be included and radomized equally to earphones with and without music.

ELIGIBILITY:
Inclusion Criteria: In the ICU, entilator treated adults > 18 years.

-

Exclusion Criteria:

* Children >18 years.
* Deaf people.
* Children <18 Years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changed dose of sedatives, | 2 times one hour
  Change of sedative treatment during mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia & Intensive Care, Karlstad, Värmland County, Sweden